CLINICAL TRIAL: NCT00656071
Title: Intraoperative Anesthetic Characteristics and the Development of ARDS
Brief Title: Retrospective Postoperative ARDS Study at Vanderbilt University
Status: Completed | Type: Observational
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Christopher Hughes, Assistant Professor, Vanderbilt University
Other Study IDs: CHughes-PGY2
Record Dates: First submitted 2008-04-04; First posted 2008-04-10 (Estimated); Last update posted 2012-09-07 (Estimated); Status verified 2012-09

CONDITIONS: ARDS
Keywords: ARDS; Acute respiratory distress syndrome; Adult respiratory distress syndrome; respiratory distress
MeSH Terms: conditions — Respiratory Distress Syndrome; Dyspnea

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Control -- postoperative mechanical ventilation patients without ARDS
- 2: Cases -- postoperative mechanical ventilation patients with ARDS

SUMMARY:
By examining the intraoperative anesthetic characteristics of patients who developed ARDS postoperatively, we hope to identify variables which have a positive or negative association on the development of ARDS.

DETAILED DESCRIPTION:
Acute respiratory distress syndrome (ARDS) is a pulmonary disease process that affects post-surgical patients in the intensive care unit and leads to significant patient morbidity and mortality and hospital cost. Extensive research has been conducted in the diagnosis and treatment of ARDS. To date, however, very little research examining the effect of the operative course on the development of ARDS has been reported. By examining the intraoperative anesthetic characteristics of patients who developed ARDS postoperatively, we hope to identify variables which have a positive or negative association on the development of ARDS. Once identified, the variables can be confirmed by future studies and encourage change in clinical care to decrease the occurrence of ARDS in surgical patients.

ELIGIBILITY:
Inclusion Criteria:

* ARDS
* post-surgical
* ventilator

Exclusion Criteria:

* rib fracture
* pneumonia
* sepsis

Min Age: 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The surgical and post-op patients at VUMC. The collection dates will be from October 1, 2001 until August 31, 2007.
Sampling Method: Non-Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2007-10; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
ARDS | data pulled from 10/2000 - 08/2007

CONTACTS AND LOCATIONS:
Overall Officials: Christopher G Hughes, M.D., Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- See also: Vanderbilt Department of Anesthesiology — http://www.vandydreamteam.com